CLINICAL TRIAL: NCT00827294
Title: A Pilot Study of Self-delivered Home-based Mirror Therapy for Phantom Limb Pain
Brief Title: Home-based Self-delivered Mirror Therapy for Phantom Limb Pain
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Beth Darnall, PhD, Associate Professor, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4925 Mirror Therapy; 5K12HD04348807
Record Dates: First submitted 2009-01-20; First posted 2009-01-22 (Estimated); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Phantom Limb Pain
Keywords: Phantom limb pain; Mirror therapy; amputation; Limb loss; treatment
MeSH Terms: conditions — Phantom Limb | interventions — Mirror Movement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Self-delivered mirror therapy (Experimental): All participants were directed to self-deliver mirror therapy for 20 minutes per day.
  Interventions: Behavioral: Mirror Therapy

INTERVENTIONS:
Behavioral: Mirror Therapy — The study is an uncontrolled pilot. Subjects receive instruction in performing mirror therapy at home, either in person or by viewing a DVD. Subjects will be asked to practice mirror therapy 20 minutes daily. Subjects will complete questionnaires for phantom pain, function, depressive symptoms, anxiety, catastrophizing, and sleep quality at baseline and post treatment at 1 month, 2 months, 3 months, and 6 months. Subjects will keep a diary of their practice and study staff will check in with subjects weekly for the first month, and monthly thereafter.

SUMMARY:
The goals of the study are to determine whether self-delivered, home-based mirror therapy decreases the frequency and intensity of phantom limb pain and improves mood and physical function in persons with phantom limb pain.

The investigators hypothesize that self-delivered home-based mirror therapy will significantly decrease phantom pain intensity, will improve mood, and will improve function at one-month follow-up.

DETAILED DESCRIPTION:
Background: Incidence of acquired amputation is increasing due to military conflict injuries and the increasing prevalence of diabetes-related peripheral vascular disease. Phantom pain is a commonly experienced comorbid condition. Existing treatments have shown mixed success in treating phantom pain. Mirror therapy has been shown to be an effective treatment when used under the guidance of a therapist in a clinical setting. There is anecdotal evidence that home-based therapy may also be effective.

Objective: Determine whether self-delivered, home-based mirror therapy decreases the frequency and intensity of phantom limb pain and improves the psychological status and physical function of amputees with phantom limb pain.

Design: Single group trial comparing pre- and post-treatment measures. Setting and Subjects: Up to 50 subjects with unilateral limb amputation and phantom limb pain will be recruited from the VA and OHSU hospital clinics. The investigators will also be passively recruiting through Kaiser Permanente Northwest (KPNW). The Pain Clinic and Physical Therapy Department at KPNW will post flyers in their waiting and patient areas for potential subjects to see. Interested patients will then self-refer to the study. Flyers will also be sent to regional amputee support groups in the Northwest and Southern California for distribution to their members. Certain inclusion and exclusion criteria must be met.

Intervention: Subjects will receive an information sheet and instruction in performing mirror therapy at home.

Measurements: Subjects will complete standard questionnaires designed to measure phantom pain level, function, depressive symptoms, pain-related anxiety, catastrophizing, and sleep quality. Subjects will also be asked about current use of pain medications and to keep a daily diary to keep track of treatment sessions.

Analysis: For the primary analysis comparing difference between baseline and 1 month post treatment, a paired t-test will be used to compare continuous variables (pain, depressive symptoms, pain-related anxiety level, sleep quality, pain catastrophizing, function) and for categorical outcomes (use of pain medications), McNemar's test or test of symmetry will be used. To investigate whether treatment gains for pain, depressive symptoms, pain-related anxiety level, sleep quality, pain catastrophizing, or function are sustained over time, a linear model will be used with controlling for correlation within repeated measures.

a. Specific Aims:

1. Primary Aim and Hypothesis: Primary Aim: Determine whether self-delivered, home-based mirror therapy decreases the intensity of phantom limb pain at one month follow-up. The primary outcome measure will be average pain intensity (the Brief Pain Inventory-short form; BPI-sf).

Hypothesis for Primary Aim #1: Amputees who practice mirror therapy at home will experience a decrease in the intensity of their phantom limb pain as measured by the Brief Pain Inventory-short form (BPI-sf) at one month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* Unilateral amputation of upper or lower limb
* At least 1 month after surgical healing
* English-speaking (since not all study materials have been translated)

Exclusion Criteria:

* History of brain injury or cognitive difficulties
* Severe mental illness that impairs cognition or function
* Suicidal ideation
* Current substance abuse or dependence
* Amputation related to diabetes

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-01; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Change in self-reported pain assessed using the Numeric Rating Scale (NRS) | month 1
  Numeric Rating Scale (NRS) ranges from score of 0 to 10, where 0=no pain and 10=worst possible pain

SECONDARY OUTCOMES:
Outcome will be determined by measuring changes in pain-related anxiety levels (baseline to one month) as measured by the Pain Anxiety Symptom Scale. | Primary interested in outcome at month 1
Change in self-reported pain assessed using the Numeric Rating Scale (NRS) | 2 months
  Numeric Rating Scale (NRS) ranges from score of 0 to 10, where 0=no pain and 10=worst possible pain

CONTACTS AND LOCATIONS:
Overall Officials: Beth D Darnall, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- [Background] Darnall BD. Self-delivered home-based mirror therapy for lower limb phantom pain. Am J Phys Med Rehabil. 2009 Jan;88(1):78-81. doi: 10.1097/PHM.0b013e318191105b. PMID 19096290